CLINICAL TRIAL: NCT06701812
Title: Evaluation of Digoxin for Relapsed Non-WNT, Non-SHH Medulloblastoma
Brief Title: Digoxin Medulloblastoma Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23221
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Medulloblastoma; Medulloblastoma, Non-WNT/Non-SHH
MeSH Terms: conditions — Medulloblastoma | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digoxin Treatment (Experimental): Digoxin will be administered orally at a standard maintenance dosing. Each cycle will be 28 days.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — 2.5-10 mcg/kg/day orally divided twice daily or once daily based on age on a continuous dosing schedule.

SUMMARY:
The purpose of this study is to evaluate the efficacy of digoxin in treating relapsed non-SHH, non-WNT medulloblastoma in pediatric and young adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age >12 months and <30 years at the time of enrollment.
* Patients must have relapsed non-WNT, non-SHH medulloblastoma confirmed by a CAP/CLIA certified assay (such as nanostring or methylation) performed on tissue from diagnosis or relapse.
* Patients must have received at least one prior course of chemotherapy for their medulloblastoma. They must also have received irradiation.
* Prior therapy: Therapy may not have been received more recently than the timeframes defined below: Craniospinal radiotherapy: At least 3 months have elapsed since prior craniospinal radiotherapy (at doses ≥ 18 Gy). Local radiotherapy: At least 3 months since prior local radiotherapy to primary tumor. Focal radiotherapy: At least 2 weeks since prior focal radiotherapy to symptomatic metastatic sites. Myelosuppressive chemotherapy and/or immunotherapy and/or biologics: More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas), immunotherapy, or biologics. Hematopoietic growth factor: Seven days must have elapsed since the completion of therapy with colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or erythropoietin), or platelet-stimulating agents.
* Patients must have recovered from any surgical procedures such as biopsy, with neurological stability for > 7 days.
* Patients must have clear residual disease, defined as tumor that is measurable in two perpendicular diameters on MRI (ie, largest tumor diameter and its largest perpendicular). The size of a measurable lesion at baseline should be at least 2 times the thickness of the slices showing the tumor (adding the interslice gap).
* Patients must have a Lansky or Karnofsky performance status score of ≥ 50%. Use Karnofsky for patients > 16 years of age and Lansky for patients < 16 years of age. Patients who are unable to ambulate but who are functional in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have normal organ and marrow function.
* Patient has no evidence of Wolff-Parkinson-White syndrome or high-grade AV block (form of second-degree heart block) on screening ECG.
* Patient has no evidence of hypertrophic obstructive cardiomyopathy on screening echo.
* Any patient that reports recent palpitations (within the last month), or concerning findings on echo or ECG must be evaluated and cleared for treatment with digoxin by a cardiologist prior to enrollment. Study PI should be contacted for additional questions/concerns regarding these patients.
* Patients receiving concurrent dexamethasone are eligible, provided dosage is stable or decreasing for ≥7 days prior to study enrollment.
* Patients must have a stable neurologic status for ≥7 days prior to study enrollment. If a patient experiences neurologic decline following enrollment but prior to day 1 of cycle 1, they should be reassessed for eligibility.
* Pregnancy: Females of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment. Female patients who are lactating must agree to stop breastfeeding.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* All patients and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent or assent document.

Exclusion Criteria:

* Participants who are receiving concurrent anticancer or any other investigational agents are ineligible.
* Participants taking digoxin for any reason during treatment for initial diagnosis of medulloblastoma or relapse are ineligible. Exposure to digoxin therapy prior to initial diagnosis of medulloblastoma is allowed.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to digoxin are ineligible.
* Patients with serious or inadequately controlled cardiac arrhythmias, including baseline ectopy, ventricular tachycardia, frequent premature ventricular contractions (PVCs), or symptomatic sinus bradycardia are excluded from the study.
* Patients taking medications that are known to interfere with digoxin metabolism are ineligible.
* Participants with uncontrolled intercurrent illness, concurrent clinically significant unrelated systemic illness (e.g. serious infection) or significant cardiac, pulmonary, hepatic, or other organ dysfunction that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results are ineligible.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements are ineligible.
* Pregnant women or women unwilling to stop breastfeeding are excluded from this study because it is unknown how pregnant women with recurrent medulloblastoma will metabolize and tolerate digoxin. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with digoxin in this setting.
* Participants who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 4 months (PFS4) | 4 months
  Proportion of patients with progression free survival at 4 months after initiation of treatment.

SECONDARY OUTCOMES:
Response rate | 4 months
  Response rate is defined as complete response (CR) + partial response (PR) at 4 months after initiation of study treatment.
Stable Disease (SD) | 4 months
  Stable disease rate as defined as stable disease (SD) at 4 months after initiation of study treatment.
Event Free Survival | Up to 12 months
  Event Free Survival as defined as time from first dose of protocol therapy to secondary malignancy, death, or progression, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Metrock, MD, Principal Investigator — University of Alabama at Birmingham Children's of Alabama; Jonathan Metts, MD, Study Chair — Moffitt Cancer Center
Locations (15):
- United States (15):
  - University of Alabama at Birmingham Children's of Alabama, Birmingham, Alabama
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Johns Hopkins All Children's, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University St. Louis, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas